CLINICAL TRIAL: NCT03495739
Title: A Randomized, Open-label, Single-dosing, 2x2 Crossover Study to Compare the Safety and Pharmacokinetics of RDG-17012(Dabigatran Etexilate Tosylate) With Pradaxa® Capsule(Dabigatran Etexilate Mesylate) in Healthy Male Volunteers
Brief Title: Clinical Trial to Assess the Safety and Pharmacokinetics of RDG-17012 Capsule and Pradaxa® Capsule in Healthy Male Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Huons Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HUG171
Record Dates: First submitted 2018-03-19; First posted 2018-04-12 (Actual); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Healthy
MeSH Terms: interventions — Dabigatran

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RDG-17012® capsule (Experimental): RDG-17012 ® capsule(dabigatran etexilate tosylate)
  Interventions: Drug: RDG-17012 Capsule
- Pradaxa® capsule (Active Comparator): Pradaxa® capsule(dabigatran etexilate mesylate)
  Interventions: Drug: Dabigatran Etexilate Mesylate 150 MG Oral Capsule

INTERVENTIONS:
Drug: RDG-17012 Capsule — Dabigatran Etexilate tosylate 150mg
  Arms: RDG-17012® capsule
Drug: Dabigatran Etexilate Mesylate 150 MG Oral Capsule — Dabigatran Etexilate mesylate 150mg
  Arms: Pradaxa® capsule

SUMMARY:
A randomized, open-label, single-dosing, 2x2 crossover study, the safety and pharmacokinetics of RDG-17012 with Pradaxa® in healthy male volunteers

ELIGIBILITY:
Inclusion Criteria:

* Age between 19 to 45, healthy male subjects(at screening)
* Subject without a hereditary problems, chronic disease and morbid symptom
* Volunteer who totally understands the progress of this clinical trials, make decision by his free will, and signed a consent form to follow the progress

Exclusion Criteria:

* Volunteer who has past or present history of any diseases following below.(liver, kidney,digestive system, pulmonary,hematooncology, endocrine, urinary,neurology,mental disorder, skeletomuscular, immunology, otolaryngology,cardiovascular)
* Exceed 2 times the normal range of AST, ALT, Total Bilirubin at screening test
* History of drug abuse, or a positive urine drug screen
* Regular alcohol consumption(over 21 units/week, 1unit=10g of pure alcohol) or volunteers who cannot abstain from drinking during the study
* Any condition that, in the view of the investigator, would interfere with study participation

Min Age: 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-06-01 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
Area Under Curve(AUC) last of Total dabigatran and Free dabigatran | (Day0)0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12hour, Day 1, Day2
Maximum of concentration(Cmax) of Total dabigatran and Free dabigatran | (Day0)0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12hour, Day 1, Day2

SECONDARY OUTCOMES:
Area Under Curve(AUC)inf of Total dabigatran and Free dabigatran | (Day0)0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12hour, Day 1, Day2

CONTACTS AND LOCATIONS:
Locations (1):
- Huons, Gyeonggi-do, Seongnam-si, South Korea

IPD SHARING:
Plan to Share IPD: No